CLINICAL TRIAL: NCT04420052
Title: Effects of Osteopathic Manipulative Treatment in Chronic Non-allergic Rhinosinusitis: a Randomised Placebo-controlled Trial
Brief Title: Effects of Osteopathic Manipulative Treatment in Chronic Non-allergic Rhinosinusitis
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: COVID, death of investigator
Sponsor: Institut des Hautes Etudes Osteopathiques de Nantes (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: Osteonose; 2019-A02907-50 (Other: Agence nationale de sécurité du médicament et produits de santé)
Record Dates: First submitted 2020-05-28; First posted 2020-06-09 (Actual); Last update posted 2023-08-01 (Actual); Status verified 2023-07

CONDITIONS: Rhinosinusitis Chronic
Keywords: Osteopathic manipulative treatment; Non-allergic; rhinosinusitis; Chronic Disease; rhinitis; sinusitis; manual therapy; osteopathy; light touch
MeSH Terms: conditions — Rhinosinusitis; Chronic Disease; Rhinitis; Sinusitis | interventions — Manipulation, Osteopathic

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Masking Description: The care provider knows the assignment of patient. In order to know if the blinding was effective, at the end of each treatment, patient will have to tell if they were in the placebo or the OMT group
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- OMT group (Experimental)
  Interventions: Other: Osteopathic manipulative treatment
- Placebo group (Placebo Comparator)
  Interventions: Other: Placebo manipulation

INTERVENTIONS:
Other: Osteopathic manipulative treatment — Osteopaths will executed several high velocity low amplitude (HVLA) techniques on the upper thoracic spine and cervical spine. These techniques are assumed to modulate the sympathetic cervical ganglia and reduce inflammation in chronic rhinosinusitis.
  This procedure takes around 15 minutes.
  Arms: OMT group
Other: Placebo manipulation — The osteopath will lay hands without movement on the nose, the throat and the thorax of patients.
  This procedure takes around 15 minutes.
  Arms: Placebo group

SUMMARY:
Chronic Rhinosinusitis (CRS) is a chronic condition with limited therapeutic options. Moreover, the pathophysiology is poorly understood. The aim of this study is to evaluate the efficacy of osteopathic manipulative treatment (OMT) in the course of this condition by applying several techniques supposed to be related to the autonomic nervous system. Our hypothesis is that these techniques could have beneficial effects on inflammation and head symptoms in CRS.

Methods:

A sample of 90 patients diagnosed by ENT specialist will be randomly assigned to the OMT group or the placebo group. The placebo procedure will consist in using light touch around the nose, on the throat and on the thorax. Treatment and placebo protocols are composed of two visits at day 0 and day 30.

A general practitioner will determine the eligibility for the study.

The outcomes include Peak Nasal Inspiratory Flow (PNIF) measured five times: at day 0, 30 (twice each, before and after treatment) and 180 (once). The two groups will be compared regarding short and long term evolution.

The evolution of symptoms will be assessed by the Sino-nasal Outcome Test (SNOT-22) seven times: at day 0, 30, 60, 90, 120, 150 and 180. This outcome will be analyzed using mixed effect modelling

A Qualitative study will be conducted in the two groups to understand the patients' experiences during care.

This protocol has been approved by a french ethic committee (Comité de Protection des Personnes Sud Ouest et Outre-Mer II, 2020.04.09).

DETAILED DESCRIPTION:
Statistical analysis details:

PNIF middle term evolution:

If the two groups can be compared regarding their socio-demographics characteristics, a student's t-test will compare evolution (day 0 before treatment to day 30 before treatment) of the PNIF between groups.

If characteristics are different, a multivariate linear model will be applied.

PNIF long term evolution:

The same tests will be made. The evolution will be assessed between day 0 (before treatment) and day 180.

PNIF short term evolution:

The same tests will be made. The evolution will be assessed before and after treatment at day 0 and day 30.

SNOT-22 evolution:

Mixed effect model will assess the evolution of symptoms from day 0 to day 180

Response Shift detection:

For the SNOT-22, an Oort procedure will be performed in order to detect Response shift among individuals.

ELIGIBILITY:
Inclusion Criteria:

* age between 18 and 50
* Chronic rhinosinusitis diagnosed by ear, nose, and throat (ENT) specialist or general practitioner
* informed consent given
* registered under french social security system

Exclusion Criteria:

* contraindication to spine manipulation
* receiving other treatment for CRS during this study
* being pregnant
* being under legal protection
* withdrawal of consent

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 0 (Actual)
Dates: Start 2021-07-01 (Estimated); Primary Completion 2022-06-01 (Estimated); Study Completion 2022-06-30 (Estimated)

PRIMARY OUTCOMES:
Change in peak nasal inspiratory flow (PNIF) | PNIF will be perform at day 0 (before treatment) and at day 30 (before treatment)
  The aim of this outcome is to measure change in nasal airflow during maximal inspiration with a facial mask.

SECONDARY OUTCOMES:
Change in Sino-nasal Outcomes Test 22 (SNOT-22) | Patients will complete the questionnaire at baseline (day 0), day 30, day 60, day 90, day 120, day 150 and day 180 to assess the change over time
  This is a symptom-based rhinosinusitis questionnaire. Possible total scores range from 0 to 110, where a higher score indicates worse symptoms.
Patient-reported experience of care | Interview will occur at day 180
  Individual interviews will enable to document the personal experience during effective or placebo treatment.
Sort term change in peak nasal inspiratory flow (PNIF) | PNIF will be perform at day 0 (before and after treatment), day 30 (before and after treatment)
  The aim of this outcome is to measure change before and after each treatment in nasal airflow during maximal inspiration with a facial mask.
long term change in peak nasal inspiratory flow (PNIF) | PNIF will be perform at day 0 (before treatment) and at day 180.
  The aim of this outcome is to measure change in nasal airflow during maximal inspiration with a facial mask from base line to day 180.

CONTACTS AND LOCATIONS:
Overall Officials: sebastien cambier, Principal Investigator — Institut des Hautes Etudes Osteopathiques de Nantes; maxime salmon, MsC, Study Director — Institut des Hautes Etudes Osteopathiques de Nantes; Marie Moreau, Study Chair — Institut des Hautes Etudes Osteopathiques de Nantes
Locations (1):
- Cabinet ORL du Maine, Le Mans, France